CLINICAL TRIAL: NCT02925611
Title: Comparison of Postoperative Delirium in Patients Anaesthetised With Isoflurane and Desflurane During Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, steve joys, Doctor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10313/PG-2Trg/2015/5408-9
Record Dates: First submitted 2016-08-27; First posted 2016-10-06 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; spine surgery; isoflurane; desflurane
MeSH Terms: conditions — Emergence Delirium | interventions — Isoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoflurane (Active Comparator): Isoflurane as an inhalational anaesthetic ,titrated with BIS ( bispectral index) /entropy monitoring,from start to end of surgery.
  Interventions: Drug: Isoflurane
- Desflurane (Active Comparator): Desflurane as an inhalational anaesthetic ,titrated with BIS ( bispectral index) /entropy monitoring,from start to end of surgery.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Isoflurane
  Arms: Isoflurane
Drug: Desflurane
  Arms: Desflurane

SUMMARY:
Postoperative delirium (POD) is a known complication of inhalational agents used to anaesthetise patients for surgery with potential long term implications.The incidence of postoperative delirium in spine surgery is 3.3% to 3.8%.The purpose of this study is to compare the occurrence of postoperative delirium with inhalational anaesthetics namely isoflurane and desflurane in spine surgery patients.

DETAILED DESCRIPTION:
The patient will be randomized to receive isoflurane or desflurane anaesthesia prior to surgery. All the patients involved in the study will be blinded to group allocation. Screening for preoperative cognitive dysfunction will be done using the mini-cog test which includes a three word recall test and clock drawing test.The primary outcome variable will be assessment of delirium at day one and day three following surgery. Post operative delirium will be diagnosed using the 3D- CAM(Confusion Assessment Method) which tests for four features with a series of questions. The features include 1) acute onset and fluctuating course,2) inattention,3) disorganized thinking and 4) altered level of consciousness. Diagnosis of delirium is made if features 1 and 2 and either 3 or 4 are present. Similarly the severity of postoperative delirium will be assessed on day one and day three following surgery. Severity of postoperative delirium will be assessed using the CAM-S(Confusion Assessment Method-severity)long form delirium severity score.It assesses ten features including 1) acute onset and fluctuating course,2)inattention,3)disorganized thinking , 4)altered level of consciousness, 5) disorientation, 6)memory impairment ,7)perceptual disturbances ,8)psychomotor agitation, 9)psychomotor retardation and 10) altered sleep-wake cycle. The scores range from 0 to 19.

The demographic data of the patients,type and site of surgery will be noted. Preoperative hemoglobin, serum electrolytes and blood urea will be recorded. The intraoperative factors like duration of surgery and anaesthesia,use of intravenous fluids ,blood loss, number blood units transfused and opioid use will be studied at the time of surgery. The time to emergence and extubation following the completion of surgery will be noted.

The postoperative factors like postoperative pain, nausea and vomiting, fever,hemoglobin,serum electrolytes and blood urea will be noted.

Preoperative and postoperative pain will be assessed using the numerical rating score on a scale of one to ten.

The association of various preoperative,intraoperative and postoperative factors with POD will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for spine surgery.
* Age between 18-65 years
* American Society of Anaesthesiologists (ASA) Grade I and II patients
* Patients with Glasgow Coma Scale (GCS) of 15
* Postoperative Aldrette score > 9

Exclusion Criteria:

* Cardiorespiratory disorders
* Associated cerebral disease
* Psychiatric illness
* Electrolyte and hormonal imbalance
* History of drug abuse
* Postoperative meningitis
* Administration of high dose steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Joys, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Hemant Bhagat, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 patients were enrolled in the study and underwent randomisation to receive isolfurane or desflurane anaesthesia with 30 patients in each group.No patients were lost to follow up and all patients were analysed.
Groups:
- Isoflurane: Isoflurane as an inhalational anaesthetic ,titrated with BIS ( bispectral index) /entropy monitoring,from start to end of surgery.
  Isoflurane
- Desflurane: Desflurane as an inhalational anaesthetic ,titrated with BIS ( bispectral index) /entropy monitoring,from start to end of surgery.
  Desflurane
Period: Overall Study
Arm/Group | Isoflurane | Desflurane
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoflurane | Desflurane | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.5 [27.5 to 40] | 37.5 [25.5 to 47.2] | 35.5 [26.2 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 23 | 20 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  India | 30 | 30 | 60
Education [Count of Participants; unit: Participants]
  uneducated(no formal education) | 0 | 1 | 1
  secondary education(5th to 12th grade) | 21 | 20 | 41
  graduate (university education) | 9 | 9 | 18
American society of anesthesiologists(ASA) status [Count of Participants; unit: Participants] — ASA 1- A normal, healthy patient ASA 2- Mild systemic disease.eg- smoker,social alcohol drinker, controlled diabetes mellitus /hypertension.
  Participants
    ASA 1 | 28 | 26 | 54
    ASA 2 | 2 | 4 | 6
comorbidities [Count of Participants; unit: Participants]
  None | 28 | 26 | 54
  Diabetes Mellitus | 1 | 1 | 2
  Hypertension | 1 | 1 | 2
  Diabetes Mellitus and Hypertension | 0 | 2 | 2
Habits [Count of Participants; unit: Participants]
  None | 19 | 23 | 42
  Alcohol | 4 | 6 | 10
  Smoking | 2 | 0 | 2
  Both | 5 | 1 | 6
diagnosis [Count of Participants; unit: Participants]
  Fracture | 14 | 11 | 25
  Intradural extramedullary tumour | 7 | 4 | 11
  Prolapse intervertebral disc | 8 | 11 | 19
  Others | 1 | 4 | 5
Hemoglobin level [Count of Participants; unit: Participants]
  <12 g /dl | 14 | 10 | 24
  >12 g/dl | 16 | 20 | 36
Preoperative serum potassium level [Count of Participants; unit: Participants]
  Normal serum potassium level | 29 | 27 | 56
  Hyperkalemia | 1 | 3 | 4
Preoperative serum sodium level [Count of Participants; unit: Participants]
  Hyonatremia | 4 | 1 | 5
  Normal serum sodium level | 26 | 28 | 54
  Hypernatremia | 0 | 1 | 1
Type of surgery [Count of Participants; unit: Participants]
  Laminectomy | 7 | 8 | 15
  Discectomy/Laminectomy and Discectomy | 7 | 9 | 16
  Pedicle screw fixation | 16 | 13 | 29
Nature of surgery [Count of Participants; unit: Participants]
  Non trauma | 16 | 19 | 35
  Trauma | 14 | 11 | 25
Level of surgery [Count of Participants; unit: Participants]
  Cervical | 4 | 2 | 6
  Dorsal | 7 | 6 | 13
  Dorsolumbar | 3 | 4 | 7
  Lumbar | 13 | 13 | 26
  Lumbosacral | 3 | 5 | 8
Position of patient [Count of Participants; unit: Participants]
  Prone | 26 | 29 | 55
  Supine | 2 | 1 | 3
  Lateral | 2 | 0 | 2
Duration of anaesthesia [Median (Inter-Quartile Range); unit: minutes] | 195 [140 to 258] | 185 [148.7 to 217.5] | 190 [142 to 226]
Duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 138 [97.5 to 196.2] | 138 [108.7 to 166.2] | 138 [102 to 180]
Number of episodes of intraoperative hypertension [Count of Participants; unit: Participants]
  0 episodes | 26 | 23 | 49
  1 episode | 2 | 6 | 8
  2 episodes | 2 | 0 | 2
  3 episodes | 0 | 1 | 1
Number of episodes of intraoperative hypotension [Count of Participants; unit: Participants]
  0 episodes | 21 | 22 | 43
  1 episode | 6 | 4 | 10
  >1 episode | 3 | 4 | 7
Median emergence time [Median (Inter-Quartile Range); unit: minutes] | 9.8 [6.8 to 14.2] | 7 [5 to 10] | 8.2 [5.4 to 12.8]
Median extubation time [Median (Inter-Quartile Range); unit: minutes] | 9.5 [6.9 to 17.2] | 9 [6 to 13.2] | 9.2 [6.2 to 15]
Intravenous fluids transfused [Median (Inter-Quartile Range); unit: millilitres] | 1500 [1500 to 2500] | 1700 [1000 to 2625] | 1600 [1200 to 2550]
Fentanyl dose [Median (Inter-Quartile Range); unit: micrograms] | 240 [170 to 290] | 220 [175 to 300] | 230 [170 to 295]
Blood loss during surgery [Median (Inter-Quartile Range); unit: millilitres] | 300 [200 to 400] | 300 [200 to 500] | 300 [200 to 500]
Number of blood units transfused [Count of Participants; unit: Participants]
  0 units | 27 | 27 | 54
  1 unit | 3 | 2 | 5
  2 units | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Postoperative Delirium(POD) With Isoflurane and Desflurane on Adults Undergoing Spine Surgery
Description: Number of Participants who were Postoperative Delirium Positive (POD+) or Negative (POD-) After Undergoing Spine Surgery With Isoflurane or Desflurane using the confusion assessment method questionnaire on day one following surgery.
Time Frame: 24 hours post surgery
Measure: Count of Participants; unit: Participants
Groups:
- Isoflurane: Isoflurane as an inhalational anaesthetic ,titrated with entropy monitoring,from start to end of surgery.
  Isoflurane
- Desflurane: Desflurane as an inhalational anaesthetic ,titrated with entropy monitoring,from start to end of surgery.
  Desflurane
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
Participants
  POD + | 3 | 4
  POD - | 27 | 26

2. Primary Outcome: Comparison of Postoperative Delirium With Isoflurane and Desflurane on Adults Undergoing Spine Surgery
Description: Number of Participants who were Postoperative Delirium Positive (POD+) or Negative (POD-) After Undergoing Spine Surgery With Isoflurane or Desflurane using the confusion assessment method questionnaire on day three following surgery.
Time Frame: 72 hours post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
Participants
  POD + | 2 | 0
  POD - | 28 | 30

3. Secondary Outcome: Post Operative Pain Scores With Isoflurane and Desflurane
Description: Comparison of postoperative pain scores (measured by numerical rating score) with by isoflurane and desflurane. The numerical rating score ranges from 0 to 10 (0 being no pain and 10 being maximum subjective pain).
Time Frame: 24 hours post surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
units on a scale | 3.5 [1 to 6.25] | 4.5 [2 to 7.25]

4. Secondary Outcome: Post Operative Pain Scores With Isoflurane and Desflurane
Description: as for outcome 3
Time Frame: 72 hours post surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
units on a scale | 1.5 [1 to 5] | 2.5 [1 to 5]

5. Secondary Outcome: CAM-S Delirium Severity Score With Isoflurane and Desflurane
Description: Comparison of CAM-S delirium severity score with isoflurane and desflurane. CAM-S delirium severity score ranges from 0 to 19 ( 0 being best outcome and 19 being worst outcome).
Time Frame: 24 hours post surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
units on a scale | 1.5 [0.75 to 4.25] | 1 [0 to 2.5]

6. Secondary Outcome: CAM-S Delirium Severity Score With Isoflurane and Desflurane
Description: as for outcome 5
Time Frame: 72 hours post surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Isoflurane | Desflurane
Number analyzed (Participants) | 30 | 30
units on a scale | 0.5 [0 to 2] | 0.5 [0 to 1]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Isoflurane | Desflurane
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
1. Small sample size
2. Postoperative delirium was assessed only up to to 72 hours post surgery. POD can persist for months following surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02925611/Prot_SAP_ICF_000.pdf